CLINICAL TRIAL: NCT01474005
Title: Establishment of an Artificial Larynx After Total Laryngectomy
Acronym: LA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4493
Record Dates: First submitted 2011-10-20; First posted 2011-11-17 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Carcinomatous Disease
Keywords: laryngectomy; artificial larynx; breathing; swallowing; upper airway
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PROTIP MEDICAL ( Artificial larynx prosthesis) — establishment of an artificial larynx prosthesis

SUMMARY:
This study aims to evaluate the effectiveness of an artificial larynx on the restoration of laryngeal functions, mainly breathing and swallowing.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over 18 years, male or female, with a carcinomatous disease of the upper airways requiring a total laryngectomy

Exclusion Criteria:

* Less than 18 years
* Contraindications to general anesthesia
* Any situation considered by the physician operator as an exclusion
* Pregnant women
* Lactating women
* Subglottic or basi-lingual tumor extension more than 1 cm
* Prior radiotherapy
* Severe coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the restoration of respiratory functions | one year
  4 items will be used:
  * 0: no dyspnea
  * 1: moderate dyspnea
  * 2: significant dyspnea
  * 3: major dyspnea
Evaluation of the restoration of the ability to swallow by nasofibroscopy | one year
  3 items will be used:
  * 1: no aspiration
  * 2: moderate aspiration
  * 3: massive aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, 1 avenue Molière, Strasbourg, France